CLINICAL TRIAL: NCT07341763
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study to Evaluate Non-invasive Brain Stimulation Effects on Orientation and Mobility Performance in Adults With Visual Impairments
Brief Title: Brain Stimulation Effects on Orientation and Mobility Skills in Adults With Vision Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: University of Waterloo School of Optometry and Vision Science (Unknown); The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Ben Thompson, Director and Professor, School of Optometry and Vision Science., University of Waterloo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB #47153
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa (RP); Rod Cone Dystrophy; Visually Impaired Persons; Peripheral Visual Field Defect of Both Eyes; Low Vision, Both Eyes; Vision Loss Partial; Orientation; Mobility Difficulty; Mobility Limitation; Mobility and Independence; Glaucoma
Keywords: Retinitis Pigmentosa (RP); Rod Cone dystrophy; Advanced Glaucoma; Visually Impaired Persons; Peripheral Visual Field Defect of Both Eyes; Low Vision, Both eyes; Brain stimulation; tES; tRNS; hf-tRNS; transcranial electrical stimulation; transcranial random noise stimulation; high-frequency transcranial random noise stimulation; Long white cane; white cane; mobility cane; walking; orientation and mobility; orientation; mobility; low vision; vision loss partial; occipital pole; primary visual cortex; V1; neuroplasticity; mobility difficulty; mobility limitation; mobility and independence
MeSH Terms: conditions — Retinitis Pigmentosa; Cone-Rod Dystrophies; Vision, Low; Orientation, Spatial; Mobility Limitation; Glaucoma

STUDY DESIGN:
Intervention Model Description: The study is a randomized, double-blind, placebo-controlled pilot study. There will be two brain stimulation/intervention sessions. The participant will receive active stimulation at one session and placebo at another sessions. Intervention sessions will be separated by 48 hours. The order will be randomized so that neither the participant nor the researcher will know what the participant will receive at each session.
Who Masked: Participant, Investigator
Masking Description: Each participant will experience active brain stimulation and placebo (sham)stimulation. The participant and the researcher will be blind to which session the participant receives active brain stimulation and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active brain stimulation (study visit 2) and Placebo/Sham (study visit 3) (Other): Participants in this arm will be exposed to active stimulation for 20 minutes whilst seated quietly at treatment session 1 (study visit 2). They will then complete the orientation and mobility (O&M) course 2-minutes and 30-minutes after stimulation. It is important to note that they will also complete the course before undergoing stimulation. In addition, individuals with constricted visual fields in both eyes who use a white cane for travelling will be encouraged to use their personal cane for the course, whereas those who do not use a cane will complete the course as they naturally would for any travel paths. Forty-eight hours later the same participants in this arm will be exposed to placebo/sham stimulation (study visit 3) and except for the treatment they receive that day, the same protocol from the previous visit will be executed, and the same outcome measures evaluated. Interventions: Active hf-tRNS at treatment (study visit 2); Placebo/sham hf-tRNS (study visit 3).
  Interventions: Device: Active hf-tRNS.; Device: Placebo/sham hf-tRNS
- Placebo/sham (study visit 2) and Active brain stimulation (study visit 3) (Other): Participants in this arm will be exposed to placebo/sham stimulation for 20 minutes whilst seated quietly at treatment session 1 (study visit 2). They will then proceed to complete the orientation and mobility (O&M) course 2-minutes and 30-minutes after stimulation. It is important to note that they will also complete the course before undergoing stimulation. In addition, individuals with constricted visual fields in both eyes who use a white cane for travelling will be encouraged to use their personal cane for the course, whereas those who do not use a cane will complete the course as they naturally would for any travel paths. Forty-eight hours later the same participants in this arm will be exposed to active stimulation (study visit 3) and except for the treatment they receive that day, the same protocol from the previous visit will be executed, and the same outcome measures evaluated. Interventions: Placebo/sham hf-tRNS at treatment (study visit 2); Active hf-tRNS (study visit 3).
  Interventions: Device: Active hf-tRNS.; Device: Placebo/sham hf-tRNS

INTERVENTIONS:
Device: Active hf-tRNS. — Active hf-tRNS: A weak alternating electric current is applied to the head through two electrodes to affect the cortical excitability of the targeted cells in the brain.
  Stimulation instrument: neuroConn DC Stimulator Plus 2019 (Direct current stimulator Model number 0021, power: 1.2 W, charger: 2.9 V (maximum 160 mA)) (neurocaregroup.com), or neuroConn DC Stimulator MC 2016 (Multi-channel stimulator Model number 0028, power: 24 W, rating: 12 V (maximum 2 A)) (neurocaregroup.com).
Device: Placebo/sham hf-tRNS — Placebo/sham hf-tRNS: The tRNS machine will be used as in active stimulation, except the electrical current will not be applied.
  Stimulation instrument: neuroConn DC Stimulator Plus 2019 (Direct current stimulator Model number 0021, power: 1.2 W, charger: 2.9 V (maximum 160 mA)) (neurocaregroup.com), or neuroConn DC Stimulator MC 2016 (Multi-channel stimulator Model number 0028, power: 24 W, rating: 12 V (maximum 2 A)) (neurocaregroup.com).

SUMMARY:
This pilot clinical trial evaluates whether non-invasive brain stimulation improves the orientation and mobility (O&M) skills of individuals with constricted visual fields in both eyes. The study is composed of three visits. The first visit is meant to confirm eligibility by performing a few clinical tests. Eligible participants will then complete two additional visits, one in which the participants receive active stimulation, and one in which the participants receive placebo (sham) stimulation. Stimulation will be administered in a randomized, double-blind order. To evaluate improvement, various measures of O&M performance will be assessed on a standardized obstacle course featuring static natural and artificial obstacles at defined intervals after the intervention. The investigators hypothesize that the application of brain stimulation to region of the brain responsible for visual processing will improve the orientation and mobility skills of individuals with binocular constricted visual fields immediately following stimulation, and the results will inform the design of a future, larger-scale study.

DETAILED DESCRIPTION:
This within-subject crossover pilot study involves applying a weak focused electrical current to the head, to target areas of visual processing, more specifically the primary visual cortex (V1) within the occipital pole. The purpose of this study is to investigate the efficacy of high-frequency transcranial random noise stimulation (hf-tRNS), a safe and well-established form of brain stimulation on O&M performance of individuals with constricted visual fields in both eyes due to either retinitis pigmentosa (RP), rod-cone dystrophy, or advanced glaucoma.

Participants will be recruited from university-affiliated clinics as well as local clinical practices. After obtaining full informed consent at the first visit, participants will complete clinical tests to confirm that the eligibility criteria of the study are met. These tests include measuring the participant's corrected binocular distance and near visual acuities, binocular contrast sensitivity, binocularity, as well as peripheral visual fields. Researchers will also ensure that it safe for the participant to undergo brain stimulation using a list of contraindicators for brain stimulation interventions and verify that participants are free from physical or motor impairments as well as vestibular disorders or dysfunctions that can impact the participant's walking and balancing abilities.

During the two subsequent visits, the effects of stimulation (which lasts 20 minutes) will be studied 2 and 30 minutes after stimulation. To evaluate improvement, various measures of O&M performance will be targeted as participants complete an O&M course divided into 4 sections and composed of an array of static natural and artificial (man-made) obstacles. Participants will be instructed to walk along the various sections at a comfortable pace, safely negotiating the obstacles without touching any of the obstacles. Participants will also be told in which sections obstacles will be encounter. Static natural obstacles refer to fixed/steady/stable obstacles that are either readily found in the environment (e.g., potted plants) or form part of the architecture of the building (e.g., a pole or a sealed doorway). Artificial obstacles are made of light materials such as polystyrene, rubber foam, soft cardboard, or paper. Static natural/real obstacles will be at foot level, foot to knee height, as well as shoulder and head heights, whereas artificial obstacles will be placed either above the knee, waist, at the shoulder or head height. Individuals with constricted field loss in both eyes who use a long white cane for travelling and have received O&M training (including caning skills) from an orientation and mobility professional will be asked to complete the course with their cane. However, individuals with constricted visual field in both eyes who do not use a cane can also complete the same course.

Measures of performance include the primary outcome measure percentage preferred walking speed (PPWS), that is the walking speed of the individual who is visually impaired in an environment with obstacles expressed as a percentage of their preferred walking speed in an unobstructed path. Secondary outcome measures include: the time taken to complete each of the 4 sections of the course, the number of O&M errors, visual detection distance (VDD) (the distance at which an individual detects an obstacle in the travel path, even if it cannot be identified), and visual identification distance (VID) (the distance at which an individual can correctly identify an obstacle in the travel path).

Course section #1 will not consist of obstacles. The time taken to complete the course section, number of O&M errors, and preferred walking speed in an unobstructed path (obtained from the completion time and length of the straight, flat path) will be measured.

Course section #2 will consist of obstacles and will be an indoor space leading to a more opened space within the building. The time taken to complete the course section, number of O&M errors, and preferred walking speed in an obstructed path (obtained from the completion time and length of the path) will be measured. The percentage preferred walking speed (PPWS) will be calculated. PPWS is the preferred walking speed of the individual in course section #2 expressed as a percentage of the participant's preferred walking speed in course section #1.

Course sections #3 and #4 will be used for measuring VDD and VID. Each course will be a straight indoor corridor consisting of only one obstacle, and the obstacle will be different for each of the two sections. Moreover, course section #3 will be used as a training course for measuring VDD and VID. The time taken to complete the course section, number of O&M errors, visual detection distance (VDD), and visual identification distance (VID) will be measured in course sections #3 and #4.

It is important to note that for course sections with obstacles (course sections # 2 to 4), the location of the obstacles in each trial (pre, post 1, and post 2) will not be varied, but rather the location of the obstacles on each treatment day will be randomized. In addition, two researchers will always be with the participant at all times. One will be with the participant to provide instructions and record data; whilst the other will be ahead of the participant to make sure the path is clear, record the times, and confirm that the obstacles are still in place (when applicable), as well as videorecord the session once consent was obtained from the participant at the first visit. By videorecording the participant as the course task is completed, the researchers will be able to obtain more accurate measures of time, and the number of O&M errors.

There will be two stimulation sessions (one with active stimulation and one with placebo (the order will be randomized so that neither the participant nor the researcher will know what the subject will receive)). At the two stimulation sessions the primary and secondary outcome measures will be evaluated as the participant completes the O&M course before stimulation (O&M pretest), as well as 2 mins after stimulation (O&M post-test 1/immediately after stimulation), and 30 mins after stimulation (O&M post-test 2/30 minutes after stimulation).

The investigators hypothesize that the application of hf-tRNS to V1 will improve the orientation and mobility skills of individuals with constricted visual fields immediately following stimulation as a result of an increase in the cortical excitability of the stimulated brain cells, which consequently leads to peripheral vision and contrast sensitivity enhancements, thereby allowing the participants to safely detect objects and obstacles in the travel path. The objective of this study is to improve the fundamental visual processes of individuals with constricted visual fields using hf-tRNS. From a scientific perspective, the investigators hope to discover whether brain stimulation can serve as an additional rehabilitation tool for improving the O&M skills of individuals with constricted visual fields. Investigators expect that participants will experience temporary O&M improvements, however, there will not be any lasting improvements in O&M skills from such a single session within subject study design. If the results of this study show a positive effect, the data will be used to power a larger study. All procedures will occur at the Human Visual Neuroscience Laboratory, University of Waterloo, Ontario, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy, capacitated adults with binocular constricted visual field loss (due to either retinitis pigmentosa (RP), rod-cone dystrophy, or advanced glaucoma) resulting in functional vision losses. These individuals with visual impairments can be those who have been previously trained by an Orientation and Mobility (O&M) specialist to independently travel with the long white cane daily (since the length of the white cane and tip at the base are based on personal preference, they should be willing to use their own white cane for the study), and those who do not necessarily use a cane for travelling.
* Have binocular visual acuity or best corrected binocular visual acuity no better than 6/12 or 20/40 or +0.30 logMAR (inclusive) with no eccentric viewing, and visual fields no better than 70 degrees in total in each eye.
* Are over the age of 18 (inclusive) and has full legal capacity to provide informed consent.
* Have read and fully comprehends the information in the consent letter.
* Are willing and capable of adhering to instructions and maintaining the outlined appointment schedule.

Exclusion Criteria:

* Are involved in other recent eye-related studies, either clinical or research-related. To be eligible they would have to wait at least one week for studies not involving brain stimulation, and four weeks for studies in which they receive brain stimulation before they could participate in this study.
* Have been diagnosed with dementia or self-reported dementia with no formal diagnosis.
* Have been diagnosed with a cognitive impairment or self-reported cognitive impairment with no formal diagnosis.
* Have been diagnosed with physical or motor impairments resulting in walking and/or balancing issues or self-reported physical or motor impairments resulting in walking and/or balancing issues with no formal diagnosis.
* Have been diagnosed with vestibular disorders or dysfunctions which affects one's balance and/or mobility or self-reported vestibular disorders or dysfunctions which affects one's balance and/or mobility with no formal diagnosis.
* Are unable to follow the researcher's instructions.
* Are anticipating treatment (including ocular surgery) for any eye disease within the duration of the study.
* Have any ocular pathology in addition to retinitis pigmentosa (RP), rod-cone dystrophy, or advanced glaucoma, which can diminish their visual acuity and/or their visual field, however wearing glasses or contact lenses, as well as mild cataract of grade 2 or below is acceptable.
* Have severe hearing impairment.
* Are pregnant or trying to get pregnant.
* Fit any of the typical contraindicators for brain stimulation. See contraindicator section below.

For all participants the contraindications for brain stimulation are:

* Diagnosed with epilepsy or have previously experienced an epileptic seizure.
* Implanted medication pump or implanted electronic device, including defibrillator or pacemaker.
* Any metal implants in the head (excluding tooth fillings).
* Active electric implants anywhere in the body (especially the head region).
* On psychoactive medication for any psychiatric or neurological conditions including but not limited to depression and schizophrenia.
* Areas of sensitive skin located on the face or head, or a skin condition on the face, or regularly use medication to alleviate skin irritation on the face.
* Recurring headaches.
* Previous head injury or skull fracture or head/brain surgery.
* Heart disease, neurological condition, or a history of cardiac or neurological surgery.
* Current or historical cancerous or noncancerous brain tumor, or other abnormalities in brain structure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage preferred walking speed (PPWS) | The pre-test and post-tests will take roughly 2 hours to complete.
  * Change in Percentage preferred walking speed (PPWS (%)) before and right after (2 mins) active stimulation.
  * Change in Percentage preferred walking speed (PPWS (%)) before and 30-minutes after active stimulation.
  * Change in Percentage preferred walking speed (PPWS (%)) before and right after (2 mins) placebo/sham stimulation.
  * Change in Percentage preferred walking speed (PPWS (%)) before and 30-minutes after placebo/sham stimulation.
  * Behavioural Measure: The participant will first complete section #1, which is obstacle free. The time taken to complete the section and preferred walking speed in an unobstructed path (obtained from the completion time and length of the straight, flat path) will be measured. They will then proceed to complete section #2, which has obstacles. The time taken to complete the section, and preferred walking speed in an obstructed path will be measured. PPWS= (preferred walking speed course 1/ preferred walking speed course 2)*100.

SECONDARY OUTCOMES:
Visual detection distance (VDD) | The pre-test and post-tests will take roughly 2 hours to complete.
  * Change in Visual detection distance (VDD (m)) before and right after (2 mins) active stimulation.
  * Change in Visual detection distance (VDD (m)) before and 30-minutes after active stimulation.
  * Change in Visual detection distance (VDD (m)) before and right after (2 mins) placebo/sham stimulation.
  * Change in Visual detection distance (VDD (m)) before and 30-minutes after placebo/sham stimulation.
  * Behavioural Measure: Participants will be instructed to walk along the various sections at a comfortable pace, safely negotiating the obstacle without touching any of them. The participant will complete sections #3 and #4. Each section will be a straight indoor corridor consisting of only one obstacle. Moreover, section #3 will be used as a training course, whereas section #4 is meant to collect data. The time it takes to first detect the obstacle and the distance from the participant to the obstacle, the moment it is first detected will be measured. This distance is VDD.
Visual identification distance (VID) | The pre-test and post-tests will take roughly 2 hours to complete.
  * Change in Visual identification distance (VID (m)) before and right after (2 mins) active stimulation.
  * Change in Visual identification distance (VID (m)) before and 30-minutes after active stimulation.
  * Change in Visual identification distance (VID (m)) before and right after (2 mins) placebo/sham stimulation.
  * Change in Visual identification distance (VID (m)) before and 30-minutes after placebo/sham stimulation.
  * Behavioural Measure: Participants will be instructed to walk along the various sections at a comfortable pace, safely negotiating the obstacle without touching any of them. The participant will complete sections #3 and #4. Each section will be a straight indoor corridor consisting of one obstacle. Section #3 will be used for training, whereas section #4 is meant to collect data. The time it takes to correctly identify the obstacle just detected, and the distance from the participant to the obstacle, the moment they first identify it will be measured (VID).
Number of orientation and mobility errors. | The pre-test and post-tests will take roughly 2 hours to complete.
  * Change in number of errors (count) before and right after (2 mins) active stimulation for course section (done for each section 1, 2, 4).
  * Change in number of errors (count) before and right after 30-minutes after active stimulation for course section (done for each section 1, 2, 4).
  * Change in number of errors (count) before and right after (2 mins) placebo/sham stimulation for course section (done for each section 1, 2, 4).
  * Change in number of errors (count) before and right after 30-minutes after placebo/sham stimulation for course section (done for each section 1, 2, 4).
  Participants will be instructed to walk along the various sections at a comfortable pace, safely negotiating any obstacles which may be present without touching any of them. The researcher will carefully observe them and note the number of errors (e.g. mobility errors- bumping into objects, orientation errors-deviations to name a few). See protocol outline document for exact error definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Thompson, PhD, Principal Investigator — University of Waterloo School of Optometry and Vision Science
Locations (1):
- University of Waterloo, School of Optometry and Vision Science, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The IPD which underlie results in a publication will be made available after deidentification upon reasonable requests to the research team.
Supporting Information: Study Protocol, SAP
Time Frame: The IPD will be available upon publication, and no more than 9 months after the publication.
Access Criteria: The IPD will be shared to researchers who provide a methodologically sound proposal.

DOCUMENTS (2):
  • Study Protocol (2025-12-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT07341763/Prot_000.pdf
  • Statistical Analysis Plan (2025-12-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT07341763/SAP_001.pdf